CLINICAL TRIAL: NCT05487820
Title: Detecting Tissue Ischemia in Reconstruction Flaps by a Novel CO2 Biosensor (DIMENSION-study); An Open, Prospective, Intervention Study
Brief Title: Detecting Tissue Ischemia in Reconstruction Flaps by a Novel CO2 Biosensor (DIMENSION-study)
Acronym: DIMENSION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sensocure AS (Industry)
Responsible Party: Principal Investigator, Magne Røkkum, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIMENSION
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ischemia; Blood Circulation Disorder; Biosensing Techniques; Surgery
Keywords: Ischemia; Biosensor; Reconstructive; Surgery; Carbon dioxide; Flap
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective, interventional. Hundred-and-sixty (56) patients will receive tissue CO2 monitoring in a reconstructed flap after reconstructive flap surgery.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with reconstructed flap monitored by tissue CO2 (Experimental): Patients scheduled for reconstructive flap surgery are monitored postoperatively with IscAlert biosensor measuring local tissue CO2 and temperature in the reconstructed flap
  Interventions: Device: IscAlert

INTERVENTIONS:
Device: IscAlert — Insertion of a CO2- and temperature sensor(s) in the reconstructed flap.

SUMMARY:
The investigators will test if changes in CO2 is detected postoperatively in ischemic tissue in a reconstructed flap.

IscAlert is measuring continuously CO2 in muscular and subcutaneous tissue. IscAlert is inserted distal to the operative field into normal muscle and/or subcutaneous tissue in the reconstructed flap. Local tissue CO2 and temperature will be monitored continuously postoperatively until maximal 10 days.

If a reduced or totally obstructed blood flow appear (thrombosis), an increase in tissue CO2 and a lower local temperature will emerge rapidly as a sign of ischemia. This will be detected by the sensor which will alarm the investigators.

This will lead to assessment of the reconstructed flap and if restricted blood flow is diagnosed, a reoperation or other intervention will be performed. 56 patients will be enrolled to undergo the procedures. The IscAlert will be removed from the patient before the patient is discharged from the hospital or a maximum of 10 days (the event that occurs first). 360 devices are planned to be used in this clinical study.

DETAILED DESCRIPTION:
This is an open, prospective, interventional, single-center clinical investigation designed to examine the feasibility and safety of the IscAlert™ device in patients scheduled for reconstructive flap surgery. 56 will be enrolled to undergo the procedures using a total of 350 devices depending on the injuries. IscAlert is 0.8 mm in diameter and in vitro testing, shows stable and accurate measurements of pCO2. More than 200 animal experiments have been done with the sensor. The experiments have shown that the sensor detects ischemia (Increased CO2-measurements) in real time in the following organs and tissues: Brain, heart, liver, kidneys, pancreas, intestines, musculature and subcutaneous tissue. Sensitivity and specificity are close to 100%. The sensors are inserted into tissue by a split needle technique. The split needle is the size of a 3-gauge peripheral venous catheter. In animal studies, no complications have been detected when using the sensor. The IscAlert sensors are connected to an electronics unit that is fixed to the skin with an adhesive plaster or glue outside the sterile area. The electrical signals are redirected to a PC approved for clinical use which continuously records tissue pressures of CO2. IscAlert is inserted into normal muscle and/or subcutaneous tissue distal on the reconstructed flap to be operated at the end of surgery. The insertion is far away from the operating field. The insertion is done under sterile conditions in accordance with standard sterility criteria at the hospital. No pain during insertion will occur because of insertion is performed during general anesthesia. Also, the insertion can be compared to an intramuscular injection. Postoperatively, the IscAlert sensor will continuously monitoring tissue CO2 and temperature. If ischemia occur, for examples caused by a thrombus, an increase in tissue CO2 and a lower temperature will evolve. This will be detected by the sensor which will alarm the investigators. This will lead to assessment of the reconstructed flap and if restricted blood flow is diagnosed, a reoperation or other intervention will be performed. The IscAlert will be removed from the patient before the patient is discharged from the hospital or a maximum of 10 days (the event that occurs first). Approximately 360 devices are planned to be used in this clinical study. One of the sensors will be used as a control inserted into neighboring tissue.

The primary objective is to compare CO2-levels in the reconstructed flap in individuals who has undergone reconstructed flap surgery and investigate if CO2-level is different in patient diagnosed with obstructed blood flow vs. patients with sufficient blood flow in the reconstructed flap.

Our hypotheses are:

1. The IscAlert™ device will be able to detect the presence of ischemia in the reconstructed flap by increased pCO2 levels and decrease in tissue temperature, measured by IscAlert™.
2. By using the IscAlert™ device monitoring ischemic events, an early treatment for ischemia could lead to higher incidence of reconstructed flap survival rates, and less revision surgery caused by thrombosis.
3. No clinically significant bleeding or infection will occur using IscAlert™ in this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled for reconstructive flap surgery
* surgery
* Patients must be ≥ 18 years
* Patients must be able to give written signed informed consent

Exclusion Criteria:

• Another study interfering with current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Tissue CO2-level | 10 days
  Tissue CO2-level (kPa) during insertion period

SECONDARY OUTCOMES:
Bleeding | 10 days
  Amount of blood from insertion site (ml)
Infection | 30 days
  Infection from insertion site at the discretion of the investigator (yes or no)
Length of stay at hospital | 30 days
  Number of days from end of initial operation to primary hospital discharge + Number of days from transfer from primary hospital to discharge from secondary hospital.
Time to reduced blood flow in reconstructed flap | 30 days
  Number of days and hours from primary surgery end to obstructed blood flow is diagnosed
Number of re-operations | 30 days
  Number of reoperations caused by replant necrosis/ischemia in the reconstructed flap

OTHER OUTCOMES:
Number of pack-years | 30 days
  Smoking habit; number of pack-years by participants
Warm ischemia time | 12 hours
  Intraoperative ischemia time of the flap (minutes)
Intravenous fluid | 12 hours
  Intravenous fluid given during surgery (ml)
Vasoactive drugs | 12 hours
  Vasoactive drugs given during surgery (microgram)
Arterial CO2 level | 10 days
  Arterial blood gass analysis of CO2 during hospital stay (kPa)
Arterial PH level | 10 days
  Arterial blood gass analysis of PH during hospital stay (kPa)
Arterial lactate level | 10 days
  Arterial blood gass analysis of lactate during hospital stay (kPa)
Arterial HCO3 level | 10 days
  Arterial blood gass analysis of HCO3 during hospital stay (kPa)
End-tidal level of CO2 | 10 days
  End-tidal level of CO2 during hospital stay (kPa)
IscAlert functionality | 10 days
  Number of hours with a well-functioning sensor (giving CO2- and temperature data)
Physical examination of the reconstructed flap - capillary filling | 10 days
  Time of capillary filling (seconds)
Physical examination of the reconstructed flap - color | 10 days
  Color of reimplanted extremity (Red or Pale)
Physical examination of the reconstructed flap - SpO2 | 10 days
  SpO2 of reimplanted extremity (%)
Physical examination of the reconstructed flap - temperature | 10 days
  Temperature of reimplanted extremity (degrees Celsius)
SpO2 | 10 days
  SpO2 measured at a finger (%)
Examination of the reconstructed flap - Doppler | 10 days
  Doppler flowmeter monitoring flow velocity in vascular flap bed (mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Magne Røkkum, MD, Ph.D, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers